CLINICAL TRIAL: NCT01592227
Title: A Pharmacokinetic Study Investigating the Rate and Extent of Absorption of Paracetamol and an Adjuvant From Two Different Paracetamol Formulations.
Brief Title: A Study to Compare Two Paracetamol Formulations.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A6480791
Record Dates: First submitted 2011-11-17; First posted 2012-05-07 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: healthy volunteer; pharmacokinetics; paracetamol
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed paracetamol (Active Comparator): Marketed paracetamol
  Interventions: Drug: Marketed paracetamol
- Experimental paracetamol formulation (Experimental): Experimental formulations
  Interventions: Drug: Experimental paracetamol formulation

INTERVENTIONS:
Drug: Marketed paracetamol — Marketed paracetamol
  Arms: Marketed paracetamol
Drug: Experimental paracetamol formulation — Experimental paracetamol formulation
  Arms: Experimental paracetamol formulation

SUMMARY:
A pharmacokinetic study investigating the rate and extent of absorption of paracetamol and an adjuvant from two different paracetamol formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers aged 18-55 years with a body mass index ranging from 19-28 kilograms per square meter who have given informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence as measured by AUC and Cmax in fasted and semi-fed states | baseline to 10 hours post dose

SECONDARY OUTCOMES:
Speed of absorption in fasted and semi-fed states | baseline to 10 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services ARIZONA, Phoenix, Arizona, United States